CLINICAL TRIAL: NCT05573113
Title: Comparative Effectiveness Trial of Bowel Ultrasound and Abdominal Radiograph Versus Abdominal Radiograph Alone for Diagnosis of Necrotizing Enterocolitis
Brief Title: Comparative Effectiveness Trial for Diagnosis of Necrotizing Enterocolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other); American College of Radiology (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Pediatric Radiologist, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00002293
Record Dates: First submitted 2022-09-23; First posted 2022-10-10 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AXR Arm 1 (Active Comparator): Abdomen Radiograph
  Interventions: Diagnostic Test: Abdominal radiograph
- AXR + BUS Arm 2 (Active Comparator): Abdomen Radiograph + Bowel Ultrasound
  Interventions: Diagnostic Test: Bowel Ultrasound; Diagnostic Test: Abdominal radiograph

INTERVENTIONS:
Diagnostic Test: Bowel Ultrasound — Bowel Ultrasound
  Arms: AXR + BUS Arm 2
Diagnostic Test: Abdominal radiograph — Abdominal radiograph

SUMMARY:
The overall objective of our study is to determine the clinical usefulness of BUS for NEC evaluation in diverse NICU settings.

DETAILED DESCRIPTION:
Bowel ultrasound (BUS) for NEC evaluation is a non-invasive imaging modality that allows real-time assessment of the intestinal wall, vascular perfusion, peristalsis, and abdominal fluid. Advantages of BUS is it is non-invasive, does not have radiation, does not require special preparation before procedure, and is well tolerated even by sick preterm infants. BUS is already being used in centers that have sufficient BUS expertise as an alternative standard of care approach for evaluating NEC, but in a highly variable manner.

Standard ultrasound equipment is all that is needed for BUS. Pre-study training will be conducted for sonographers to acquire the study BUS images using standardized technique. Pre-study training of radiologists will also be conducted to standardize the interpretation of BUS findings for NEC. All BUS for NEC ordering, acquisition, and interpretation in the study will be the same as the standard workflow for any other imaging ordered in the clinical setting. All BUS performed as part of the study will not be charged to patients.

ELIGIBILITY:
Inclusion Criteria

* Admitted to the NICU at CMKC or KUMC
* With clinical suspicion for NEC for which further imaging evaluation was decided by treating neonatologist

Exclusion Criteria

• Infants with major gastrointestinal anomalies such as gastroschisis or omphalocele that prevent BUS from being performed

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Chan, MD, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted between Sept 2022 - Dec 2024 at two sites: Children's Mercy Hospital (Level IV NICU) and University of Kansas Medical Center (Level III NICU).
Pre-assignment Details: Randomization was conducted by calendar month (odd months = AXR only; even months = AXR + BUS). Cross-over occurred in 31 AXR-only evaluations (also received BUS) and 3 AXR+BUS evaluations (only received AXR). A total of 169 infants underwent 199 imaging evaluations for NEC.
Units Other Than Participants: Imaging evaluation for NEC
Groups:
- Abdominal Radiographs Only (AXR): Infants with concern for necrotizing enterocolitis randomized to imaging with abdominal radiographs only (AXR)
- Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS): Infants with concern for necrotizing enterocolitis randomized to imaging with abdominal radiographs plus bowel ultrasound (AXR + BUS)
Period: Overall Study
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Started | 92; 114 Imaging evaluation for NEC (92 infants with 114 distinct imaging evaluations for NEC concern randomized to AXR only) | 77; 85 Imaging evaluation for NEC (77 infants with 85 distinct imaging evaluations for NEC concern randomized to AXR + BUS)
Cross-Over | 26; 31 Imaging evaluation for NEC (26 infants with 31 distinct imaging evaluations for NEC concern randomized to AXR only but cross-over to AXR + BUS) | 3; 3 Imaging evaluation for NEC (3 infants with 3 distinct imaging evaluations for NEC concern randomized to AXR + BUS but cross-over to AXR only)
Completed | 92; 114 Imaging evaluation for NEC (Analysis by Intention-to-treat to preserve randomization) | 77; 85 Imaging evaluation for NEC (Analysis by intention-to-treat to preserve randomization)
Not Completed | 0; 0 Imaging evaluation for NEC | 0; 0 Imaging evaluation for NEC

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs Plus Bowel Ultrasound (AXR + BUS) | Total
Number analyzed (Participants) | 92 | 77 | 169
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 31 (4.8) | 31 (5.2) | 31 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 56
  Male | 55 | 58 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 18 | 39
  White | 46 | 40 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 15 | 37
Birthweight [Mean (Standard Deviation); unit: kg] | 1.63 (0.86) | 1.66 (1.10) | 1.64 (0.97)
Site - Level III or IV NICU [Count of Participants; unit: Participants]
  Level III | 37 | 27 | 64
  Level IV | 55 | 50 | 105
Multiple Gestation (%) [Count of Participants; unit: Participants] | 18 | 17 | 35
Congenital anomalies (%) [Count of Participants; unit: Participants] | 19 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Days to Full Enteral Feeds: Extended Rule Out Group
Description: Number of days for infants to tolerate at least 120 mL/kg/day of enteral feeds
Time Frame: Within 30 days of NEC concern
Population: Extended Rule Out Group: Infants with clinical concern for NEC who were ultimately not diagnosed with NEC but required more than one AXR to confidently rule out the disease. Infants who crossed over to a different imaging strategy were analyzed according to the arm to which they were originally randomized, following an intention-to-treat approach.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 42 | 28
days | 10.1 (10.9) | 4.9 (4.5)

2. Primary Outcome: Days to Full Enteral Feeds: Quick Rule Out Group
Description: Number of days for infants to tolerate at least 120 mL/kg/day of enteral feeds
Time Frame: Within 30 days of NEC concern
Population: Quick Rule Out Group: Infants with suspected NEC in whom the diagnosis was excluded after a single AXR. Infants who crossed over to a different imaging strategy were analyzed according to the arm to which they were originally randomized, following an intention-to-treat approach.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 40 | 23
days | 0.4 (1.4) | 1.0 (2.4)

3. Primary Outcome: Days to Full Enteral Feeds: NEC Ruled In
Description: Number of days for infants to tolerate at least 120 mL/kg/day of enteral feeds
Time Frame: Within 30 days of NEC concern
Population: NEC Ruled In Group: Infants with suspected NEC who were diagnosed with NEC based on clinical, laboratory, and imaging findings. Infants who crossed over to a different imaging strategy were analyzed according to the arm to which they were originally randomized, following an intention-to-treat approach.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 32 | 34
days | 17.0 (8.6) | 17.6 (9.0)

4. Secondary Outcome: Days to End Bowel Rest: Extended Rule Out Group
Description: Number of days infants were kept nil per os (without enteral feeds) following concern for NEC
Time Frame: within 14 days of NEC concern
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 42 | 28
days | 2.6 (2.9) | 2.1 (1.8)

5. Secondary Outcome: Days to End Bowel Rest: Quick Rule Out Group
Description: Number of days infants were kept nil per os (without enteral feeds) following concern for NEC
Time Frame: within 14 days of NEC concern
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 40 | 23
days | 0.2 (0.6) | 0.4 (0.8)

6. Secondary Outcome: Days to End Bowel Rest: NEC Ruled In
Description: Number of days infants were kept nil per os (without enteral feeds) following concern for NEC
Time Frame: within 14 days of NEC concern
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 32 | 34
days | 8.7 (4.0) | 8.7 (3.5)

7. Secondary Outcome: Days to End Antibiotics: Extended Rule Out
Description: Number of days infants received antibiotic therapy initiated for NEC concern
Time Frame: within 14 days of NEC concern
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 42 | 28
days | 1.6 (2.3) | 1.5 (2.3)

8. Secondary Outcome: Days to End Antibiotics: Quick Rule Out
Description: Number of days infants received antibiotic therapy initiated for NEC concern
Time Frame: within 14 days of NEC concern
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 40 | 23
days | 0.1 (0.8) | 0.8 (3.1)

9. Secondary Outcome: Days to End Antibiotics: NEC Rule In
Description: Number of days infants received antibiotic therapy initiated for NEC concern
Time Frame: within 14 days of NEC concern
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS)
Number analyzed (Participants) | 32 | 34
days | 8.4 (4.0) | 7.5 (3.2)

ADVERSE EVENTS:
Time Frame: Until discharge from hospital or death, up to a maximum of 180 days.
Groups:
- Cross-Over to AXR + BUS: Infants with concern for necrotizing enterocolitis randomized to imaging with abdominal radiographs only (AXR) but cross-over to AXR + BUS
- Cross-Over to AXR only: Infants with concern for necrotizing enterocolitis randomized to imaging with abdominal radiographs plus bowel ultrasound (AXR + BUS) but cross-over to AXR only
Arm/Group | Abdominal Radiographs Only (AXR) | Abdominal Radiographs plus Bowel Ultrasound (AXR + BUS) | Cross-Over to AXR + BUS | Cross-Over to AXR only
All-Cause Mortality (participants affected / at risk) | 5/66 | 8/74 | 1/26 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/74 | 0/26 | 0/3
Other Adverse Events (participants affected / at risk) | 0/66 | 0/74 | 0/26 | 0/3

LIMITATIONS AND CAVEATS:
* Cross-over between study arms occurred.
* Study conducted at only two sites; generalizability may be limited.
* Some analyses underpowered due to smaller sample size than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT05573113/Prot_SAP_001.pdf